CLINICAL TRIAL: NCT00457197
Title: Quetiapine for Bipolar Disorder and Alcohol Dependence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU 072010-090
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Results first posted 2016-01-28 (Estimated); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Bipolar Disorder; Alcohol Dependence
Keywords: bipolar disorder; alcohol dependence; mania; manic disorder; depression
MeSH Terms: conditions — Bipolar Disorder; Alcoholism; Mania; Depression | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): This group will be given placebo matching quetiapine for the course of the 12 weeks in the study.
  Interventions: Drug: Placebo
- Quetiapine (Active Comparator): This group will be given 50mg Quetiapine per day baseline-week 1, 100mg Quetiapine per day week 1-week 2, 200mg Quetiapine per day week 2-week 3, 400mg Quetiapine per day week 3-week 4, and 600mg Quetiapine per day week 4 to week 12.
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Placebo — Inactive ingredient matching the active medication in appearance.
  Other Names: Sugar-pill
  Arms: Placebo
Drug: Quetiapine — Quetiapine is an atypical antipsychotic approved for the treatment of schizophrenia, bipolar disorder, and in the XR version along with an SSRI to treat major depressive disorder.
  Other Names: Seroquel; Xeroquel; Ketipinor
  Arms: Quetiapine

SUMMARY:
The purpose of this study is to find out whether an investigational drug called quetiapine can treat bipolar disorder, improve mood and reduce alcohol use and craving.

DETAILED DESCRIPTION:
The primary aim in the study is to determine if quetiapine treatment is associated with greater reduction in alcohol use than placebo in outpatients with bipolar disorder and alcohol dependence. We will also examine if quetiapine treatment is associated with greater reduction in alcohol craving than placebo in outpatients with bipolar disorder and alcohol dependence and if quetiapine treatment is associated with greater improvement in depressive symptoms than placebo in outpatients with bipolar disorder and alcohol dependence.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with a diagnosis of bipolar I or II disorder, depressed or mixed phase on the Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders (SCID) and confirmed by interview with PI or co-I.
* Current diagnosis of alcohol dependence.
* Alcohol use (by self-report) of at least 15 drinks in the 7 days prior to baseline.
* Currently taking a mood stabilizer defined as lithium, divalproex/valproic acid, oxcarbazepine, or lamotrigine at a stable dose for > 14 days.
* Men and women age 18-65 years old.
* English or Spanish speaking.

Exclusion Criteria:

* Bipolar disorders other than bipolar I or II (e.g., not otherwise specified or cyclothymic disorders) based on the SCID and confirmed through clinical assessment by PI or co-I.
* Baseline Young Mania Rating Scale (YMRS) score > 35 or Hamilton Depression Rating Scale (HRSD) 17 score > 35.
* Current clinically significant psychotic features (hallucinations, delusions, disorganized thought processes).
* Evidence of clinically significant alcohol withdrawal symptoms defined as a Clinical Institute Withdrawal Assessment (CIWA-AR) score of > 8.
* History of hepatic cirrhosis or baseline AST or ALT > 3X upper limit of normal or other clinically significant findings on physical or laboratory examination.
* Mental retardation or other severe cognitive impairment.
* Prison or jail inmates.
* Pregnant or nursing women or women of childbearing age who will not use oral contraceptives, abstinence, or other acceptable methods of birth control during the study.
* Antipsychotic therapy within 14 days prior to randomization.
* Current carbamazepine or benzodiazepine therapy.
* Current treatment with medications shown to reduce alcohol consumption (naltrexone, acamprosate, disulfiram, or topiramate) in large randomized, controlled trials.
* Initiation of antidepressants or mood stabilizers or psychotherapy within past 2 weeks.
* High risk for suicide, defined as any suicide attempts in the past 3 months or current suicidal ideation with plan and intent.
* Intensive outpatient treatment for substance abuse (AA, NA meetings, or other 12-step programs or weekly psychotherapy that started at least 14 days prior to randomization will be allowed).
* Current treatment with ketoconazole, itraconazole, erythromycin, or nefazodone.
* Severe or life-threatening medical condition (e.g., congestive heart failure, terminal cancer) or laboratory or physical examination findings consistent with serious medical illness (e.g., severe edema, atrial fibrillation, dangerously abnormal electrolytes).
* Diabetes mellitus by history or suspected from baseline blood sugar.
* History of cataracts or suspected cataracts on ophthalmic exam
* History of seizure disorder of any etiology; if a subject develops a seizure episode, s/he will be discontinued from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2007-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Sherwood Brown, MD PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Psychoneuroendocrine Research Program, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Quetiapine
Started | 45 | 45
Completed | 44 | 44
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Quetiapine | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (10.1) | 43.3 (8.2) | 41.5 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 25 | 27 | 52
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 21 | 21 | 42
  African American | 12 | 13 | 25
  Hispanic | 10 | 7 | 17
  Other | 1 | 2 | 3
  Missing | 0 | 1 | 1
Married [Number; unit: participants]
  Married | 8 | 10 | 18
  Not Married | 36 | 34 | 70
Education [Mean (Standard Deviation); unit: years] | 13.3 (2.4) | 13.6 (2.5) | 13.5 (2.5)
Mood states [Number; unit: participants]
  Depressed | 40 | 38 | 78
  Mixed (both depression and mania at same time) | 4 | 6 | 10
History of treatment for drug/alcohol [Number; unit: participants]
  History | 25 | 30 | 55
  No History | 19 | 14 | 33
% Days Alcohol Use In Past Week [Mean (Standard Deviation); unit: days] | 74.6 (26.1) | 74.2 (27.3) | 74.4 (26.7)
% Days Heavy Alcohol Use In Past Week [Mean (Standard Deviation); unit: Days] | 60.0 (30.1) | 53.0 (30.9) | 56.5 (30.5)
Drinks per day [Mean (Standard Deviation); unit: drinks] | 6.5 (3.4) | 6.0 (3.4) | 6.3 (3.4)
Liver enzymes [Mean (Standard Deviation); unit: IU/I]
  GGT (gamma-glutamyltransferase | 47.8 (37.6) | 74.3 (69.3) | 61.05 (53.45)
  AST (aspartate aminotransferase) | 27.4 (14.8) | 29.7 (13.5) | 28.6 (14.2)
  ALT (alanine aminotransferase) | 29.0 (24.5) | 28.9 (17.3) | 29.0 (20.9)
Concomitant medications [Number; unit: participants]
  Lithium | 28 | 27 | 55
  No Lithium | 16 | 17 | 33
Concomitant medications [Number; unit: participants]
  Anticonvulsants | 13 | 13 | 26
  No anticonvulsants | 31 | 31 | 62
Concomitant medications [Number; unit: participants]
  Antidepressants | 6 | 11 | 17
  No antidepressants | 38 | 33 | 71
Concomitant medications [Number; unit: participants]
  Sedatives/hypnotics | 2 | 8 | 10
  No sedatives/hypnotics | 42 | 36 | 78
Mood and craving scales: Hamilton Rating Scale for Depression [Mean (Standard Deviation); unit: units on a scale] — Minimum: 0 Maximum: 50 Lower score associated with better outcome Normal= 7 or less
  units on a scale | 18.3 (6.7) | 18.6 (7.0) | 18.5 (6.9)
Mood and craving scales: Inventory of Depressive Symptomatology-Self-Report [Mean (Standard Deviation); unit: units on a scale] — Minimum= 0 Maximum= 84 Lower score associated with better outcome Normal= 7 or less
  units on a scale | 28.6 (10.7) | 33.9 (14.6) | 31.3 (12.65)
Mood and craving scales: Young Mania Rating Scale [Mean (Standard Deviation); unit: units on a scale] — Minimum: 0 Maximum: 60 Lower score associated with better outcome
  units on a scale | 13.6 (8.2) | 13.9 (6.7) | 13.8 (7.5)
Mood and craving scales: Penn Alcohol Craving Scale [Mean (Standard Deviation); unit: units on a scale] — Minimum: 0 Maximum: 30 Lower score associated with better outcome
  units on a scale | 19.2 (6.6) | 20.6 (6.3) | 19.9 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Standard Drinks/Day Will Serve as the Primary Outcome Measure.
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: drinks
Arm/Group | Placebo | Quetiapine
Number analyzed (Participants) | 44 | 44
drinks | 10.6 (2.465) | 8.09 (2.465)
Statistical Analysis 1: Comparison: Placebo vs Quetiapine; Baseline drinks/day used as covariate; Test type: Superiority or Other; p = 0.4709, ANCOVA

2. Secondary Outcome: Percent of Heavy Drinking Days
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: drinks
Arm/Group | Placebo | Quetiapine
Number analyzed (Participants) | 44 | 44
drinks | 28.8 (3.66) | 20.8 (3.66)
Statistical Analysis 1: Comparison: Placebo vs Quetiapine; Baseline percent heavy drinking days included as covariate; Test type: Superiority or Other; p = 0.1272, ANCOVA

3. Secondary Outcome: Gamma-glutamyltransferase (GGT)
Description: GGT is a liver enzyme measurement (IU/I)
Time Frame: 12 weeks
Population: Missing data for 18 participants in placebo group and 11 participants in the quetiapine group.
Measure: Least Squares Mean (Standard Error); unit: IU/I
Arm/Group | Placebo | Quetiapine
Number analyzed (Participants) | 26 | 33
IU/I | 66.6 (8.34) | 66.0 (7.38)
Statistical Analysis 1: Comparison: Placebo vs Quetiapine; Baseline GGT used as covariate; Test type: Superiority or Other; p = 0.9642, ANCOVA

4. Secondary Outcome: Aspartate Aminotransferase (AST)
Description: AST is a liver enzyme measurement (IU/I)
Time Frame: 12 weeks
Population: Missing data for 19 participants in placebo group and 11 participants in the quetiapine group.
Measure: Least Squares Mean (Standard Error); unit: IU/I
Arm/Group | Placebo | Quetiapine
Number analyzed (Participants) | 25 | 33
IU/I | 29.7 (2.92) | 31.1 (2.54)
Statistical Analysis 1: Comparison: Placebo vs Quetiapine; Baseline AST used as covariate; Test type: Superiority or Other; p = 0.7222, ANCOVA

5. Secondary Outcome: Alanine Aminotransferase (ALT)
Description: ALT is a liver enzyme measurement (IU/I).
Time Frame: 12 weeks
Population: Missing data for 17 participants in placebo group and 13 participants in the quetiapine group.
Measure: Least Squares Mean (Standard Error); unit: IU/I
Arm/Group | Placebo | Quetiapine
Number analyzed (Participants) | 27 | 31
IU/I | 25.1 (2.61) | 30.4 (2.43)
Statistical Analysis 1: Comparison: Placebo vs Quetiapine; Baseline ALT used as covariate; Test type: Superiority or Other; p = 0.1412, ANCOVA

6. Secondary Outcome: Hamilton Rating Scale for Depression (HRSD)
Description: The assessment is a clinician administered rating of depression with 17 questions. The total score is indicates level of depression within the following ranges: none (0-5), mild (6-10), moderate (11-15), severe (16-20), and very severe (21+).
  Scale:
  Minimum: 0 Maximum: 50 Lower score associated with better outcome
Time Frame: 12 weeks
Population: Missing data for 2 participants in placebo group and 3 participants in the quetiapine group.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Quetiapine
Number analyzed (Participants) | 42 | 41
units on a scale | 10.9 (1.10) | 10.3 (1.12)
Statistical Analysis 1: Comparison: Placebo vs Quetiapine; Baseline HRSD used as covariate; Test type: Superiority or Other; p = 0.7071, ANCOVA

7. Secondary Outcome: Inventory of Depressive Symptomatology-Self Report (IDS-SR)
Description: IDS-SR is a self reported 30 item assessment to diagnose a major depressive episode.
  Score:
  Minimum: 0 Maximum: 84 Lower score associated with better outcome
Time Frame: 12 weeks
Population: Missing data for 4 participants in placebo group and 2 participants in the quetiapine group.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Quetiapine
Number analyzed (Participants) | 40 | 42
units on a scale | 19.0 (1.79) | 21.9 (1.75)
Statistical Analysis 1: Comparison: Placebo vs Quetiapine; Baseline IDS-SR used as a covariate; Test type: Superiority or Other; p = 0.2569, ANCOVA

8. Secondary Outcome: Young Mania Rating Scale (YMRS)
Description: This is an 11-item, observer rated measure of the severity of manic symptoms on a 5 point scale. The total score indicates overall severity of mania with a minimum of zero (indicating normalcy) and a maximum of 60 (indicating very severe).
  Score:
  Minimum: 0 Maximum: 60 Lower score associated with better outcome
Time Frame: 12 weeks
Population: Missing data for 6 participants in placebo group and 1 participant in the quetiapine group.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Quetiapine
Number analyzed (Participants) | 38 | 43
units on a scale | 8.70 (1.09) | 8.48 (1.02)
Statistical Analysis 1: Comparison: Placebo vs Quetiapine; Baseline YMRS used as a covariate; Test type: Superiority or Other; p = 0.8814, ANCOVA

9. Secondary Outcome: Penn Alcohol Craving Scale (PACS)
Description: The PACS is a five-item self-administered instrument for assessing craving, frequency, intensity, and duration of thoughts about drinking are assessed along with ability to resist drinking
  Score:
  Minimum: 0 Maximum: 30 Lower score associated with better outcome.
Time Frame: 12 weeks
Population: Missing data for 1 participants in placebo group and 5 participants in the quetiapine group.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Quetiapine
Number analyzed (Participants) | 43 | 39
units on a scale | 14.1 (1.03) | 12.3 (1.09)
Statistical Analysis 1: Comparison: Placebo vs Quetiapine; Baseline PACS used as a covariate; Test type: Superiority or Other; p = 0.2473, ANCOVA

ADVERSE EVENTS:
Arm/Group | Placebo | Quetiapine
Serious Adverse Events (participants affected / at risk) | 3/45 | 5/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=45) | Quetiapine (N=45)
Myocardial Infarction (Cardiac disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Victim of Sexual Assault (Injury, poisoning and procedural complications) | 0 | 1
Arrest for Public Intoxication (Psychiatric disorders) | 1 | 1
Panic Attack (Psychiatric disorders) | 0 | 1
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Larger sample size possibly needed for between-group differences in outcome measures. Pill counts not an optimum measure of medication adherence.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No